CLINICAL TRIAL: NCT04272528
Title: Construction and Evaluation of a Uniform Stoma Patient Care Network in Shaanxi Province
Brief Title: Construction and Evaluation of a Stoma Patient Care Network
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019SF-124
Record Dates: First submitted 2019-12-30; First posted 2020-02-17 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Surgical Stomas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Nurses provide uniform care to patients according to the quality standards.
  Interventions: Other: uniform care
- control group (Placebo Comparator): Nurses provide the routine care to patients.
  Interventions: Other: conventional care

INTERVENTIONS:
Other: uniform care — The leader develops training plan and trains nurses, who provide uniform care and education to patients according to the training.
  Arms: experimental group
Other: conventional care — Nurses carry out the routine care procedures.
  Arms: control group

SUMMARY:
Establish a uniform care network for stoma patients in Shaanxi Province and evaluate its effectiveness, so that stoma patients can get the same quality of stoma care outside the hospital.

DETAILED DESCRIPTION:
This project plans to take the First Affiliated Hospital of Xi'an Jiaotong University as the lead hospital to establish a uniform care network for stoma patients in Shaanxi Province. This network includes the management system of stoma nursing and the management organization of stoma patients in Shaanxi Province. It formulates the whole quality standard of stoma nursing in Shaanxi Province, carries out "standard training" for the stoma specialty nurses in the group, and carries out on-site inspection in various hospitals from time to time, establishes the feedback mechanism and standardizes the stoma nursing process. The contact card of stoma therapists was made and distributed to patients with stoma, so that patients can easily get the information of stoma therapists in the nearest hospital and receive professional and convenient care. WeChat group of specialized stoma nurses was established to provide remote guidance for difficult cases, share new stoma ideas and knowledge, and facilitate communication among stoma nurses in the group. The leading hospital holds training courses on knowledge and progress of stomatology every year, competitions on knowledge and skills, and dispatches therapists to provide work guidance, so as to share new knowledge, skills and scientific research abilities. At the same time, the efficacy of the network was evaluated by investigating the complication rate, self-care ability, quality of life, medical costs of stoma patients,as well as the specialized nursing skills and professional development of nurses.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥18 years old;
* patients undergoing enterostomy;
* patients with primary school and above education level;
* patients with clear consciousness, reading and verbal expression ability;
* patients could reexamine regularly;
* patients informed consent and voluntary participation in the study.

Exclusion Criteria:

* patients with organ dysfunction who have difficulty in self-care;
* patients with mental illness, consciousness disorder or communication disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life measured by Stoma Quality of Life (Stoma-QOL). | 6 months
  The scale includes 20 items with a score ranging from 20 to 80 points. The higher the score, the better the quality of life.

SECONDARY OUTCOMES:
Self-care ability measured by stoma self-care ability scale | 6 months
  The scale includes three dimensions: self intention questionnaire (12-48 points), self-care knowledge (0-21 points), self-care skills (0-12 points). The higher the score, the higher the self-care ability.
Stoma complications | 6 months
  Stoma complications include infection around the stoma，parastomal hernia，skin and mucous membrane separation，fistula of stoma，hemorrhage，ischemia，and stenosis．

CONTACTS AND LOCATIONS:
Overall Officials: Xia Xin, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No